CLINICAL TRIAL: NCT05518201
Title: Evaluate the Safety and Immunogenicity of the 9-valent Human Papillomavirus Recombinant Vaccine (Hansenula Polymorpha) in Chinese Male Aged 9-45 Years: A Randomized, Blinded and Placebo-Controlled Phase I Study
Brief Title: Evaluate the Safety and Immunogenicity of a 9-valent HPV Vaccine in Chinese Healthy Male Aged 9-45 Year-old
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Bovax Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 9-HPV-1002
Record Dates: First submitted 2022-08-25; First posted 2022-08-26 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2022-10

CONDITIONS: Penile Cancer; Anal Cancer; PIN-1; PIN-2; PIN-3; AIN1; AIN2; AIN3; Genital Wart
MeSH Terms: conditions — Penile Neoplasms; Anus Neoplasms; Condylomata Acuminata

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The 9vHPV Recombinant Vaccine among 18-45yrs (Experimental): Subjects received 3 doses of 9-valent HPV vaccine according to a 0, 2, 6-month schedule (0.5mL/each dose).
  Interventions: Biological: Placebo among 18-45 yrs
- The 9vHPV Recombinant Vaccine among 9-17 yrs (Experimental): Subjects received 3 doses of 9-valent HPV vaccine according to a 0, 2, 6-month schedule (0.5mL/each dose).
  Interventions: Biological: Placebo among 9-17 yrs

INTERVENTIONS:
Biological: Placebo among 18-45 yrs — Subjects received 3 doses of placebo according to a 0, 2, 6-month schedule (0.5mL/each dose).
  Arms: The 9vHPV Recombinant Vaccine among 18-45yrs
Biological: Placebo among 9-17 yrs — Subjects received 3 doses of placebo according to a 0, 2, 6-month schedule (0.5mL/each dose).
  Arms: The 9vHPV Recombinant Vaccine among 9-17 yrs

SUMMARY:
To evaluate the safety and tolerability of the 9vHPV vaccine in Chinese healthy male aged 9 to 45 years.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Chinese male aged 9 to 45 years; Provide legal identification; For those under the age of 18, they must also provide their guardian's legal identification;
2. Adults voluntarily agrees to enroll in this study. If the subject is a minor, both the subject and subject's legal guardian should voluntarily agree to enroll in this study and sign an informed consent form;
3. Subjects and/or their legal guardian are able to read and understand the study schedule, and commitment to regular follow-up as required by the study;
4. Subjects will take effective contraception from Day 0 to month 7 (For Male: celibate, wear a condom, vasectomy, etc. ; For Female Sexual Partners: use IUD, oral/injecting/Slow-release topical contraceptives (except emergency contraceptives), Hormone patches, sterilization, contraceptive diaphragm, etc.

Exclusion Criteria:

1. Subjects aged over 14 years on the day of enrolment had fever (axillary temperature≥37.3℃) within 24 hours prior to the first dose of vaccination; subjects aged≤14 had fever within 24 hours prior to the first dose of vaccination (axillary temperature≥37.5℃);
2. Poor controlled hypertension, i.e., after lifestyle modification and/or treated (aged 9 to 17 years: systolic BP≥120mmHg and/or diastolic BP≥80mmHg; aged 18 to 45 years: Systolic BP≥140mmHg and/or diastolic BP ≥90mmHg);
3. Had received marketed HPV vaccine; plan to receive marketed HPV vaccine during this study period; have enrolled in HPV vaccine clinical trials and have received trial vaccine/placebo;
4. History of positive test to HPV (including types not covered by 9vHPV vaccine);
5. History of external genital disease (e.g. genital warts, penis/perianal region/perineum intraepithelial neoplasia, penile/perianal/perineal cancer), diseases within the anus (e.g. anal intraepithelial neoplasia and anal cancer), or history of head and neck cancer;
6. Present history of severe liver and kidney disease, severe CVDs, severe hypertension, diabetic complications, or history of malignant tumour;
7. History of convulsions (except fever convulsions in children under 2 years of age), epilepsy, brain diseases, mental illness, or family history;
8. With prohibitive contraindications to intramuscular injection, such as Thrombocytopenia, coagulopathy, or being treated with anticoagulants;
9. Asplenic, functionally asplenic, or splenectomy caused by any condition;
10. History of severe allergic reactions requiring medical intervention (e.g., anaphylactic shock, allergic laryngeal edema, Anaphylactoid purpura, thrombocytopenic purpura, local allergic necrosis reaction (Arthus reaction), etc.); History of severe side effects or a history of severe allergies to any of the components of the vaccine (Histidine, Polysorbate 80, Aluminum Phosphate Adjuvant);
11. History of congenital/acquired immunodeficiency, such as lymphoma, leukemia, systemic lupus erythematosus, rheumatoid arthritis, juvenile rheumatoid arthritis, Inflammatory bowel disease, or other autoimmune diseases, etc.; Received immunosuppressive treatment within 6 months before vaccination, such as long-term glucocorticoid use (Dosage reference: equivalent to prednisone 20mg per day, more than one week); Or monoclonal antibodies; Or thymus peptides; Or interferon, etc.; Or plan to receive such products during this study period (From Day 0 to Month 7); Allow topical medication (e.g., ointments, eye drops, inhalants, or nasal sprays, etc.);
12. Present history of infectious diseases, such as Tuberculosis (TB), Hepatitis, HIV infection, and/or TeponemaPllidum infection;
13. Within 3 days prior to vaccination, have an acute disease or are in the acute attack of a chronic disease or have used antipyretic, analgesic and anti-allergic drugs (such as: acetaminophen, ibuprofen, aspirin, loratadine, cetirizine, etc.);
14. Inactivated/recombinant/nucleic acid vaccines, etc. (non-attenuated vaccines) have been given within 14 days before enrollment; or have been vaccinated within 28 days of attenuated vaccines; or have received immunoglobulin products or blood-related products within 3 months before enrollment;
15. Received other investigative or unregistered products within 30 days before vaccination or plan to receive such products during this study period; Or still participating in other clinical trial within 3 months prior to enroll this study;
16. Plan to receive immunoglobulin products or blood-related products during this study period (From Day 0 to Month 7);
17. Plan to relocate permanently from the area before the end of the study or leave the local area for a long time during the study visit (affecting the scheduled visit time);
18. Abnormal laboratory testing indicators specified in study protocol (except NCS);
19. According to the investigator's judgment, the subjects had any condition that were not suitable for participation in this study.

Ages: 9 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Adverse Events (AEs) | From Day 0 to Month 7
  Subjects with solicited and unsolicited AEs
Number of subjects with Severe adverse events (SAE) | From Day 0 to Month 12
  SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects.

SECONDARY OUTCOMES:
Number of subjects receiving the 3-doses scheduled vaccination with antibody responses as assessed by Geometric mean titer (GMT) | day 31 post last dose
  Immunogenicity were assessed by the GMT of anti HPV6/11/16/18/33/45/52/58 neutralizing antibodies after day 31 post last dose, among the subjects who were aged 9-45
Number of subjects receiving the 3-doses scheduled vaccination with antibody responses as assessed by seroconversion rate | day 31 post last dose
  Immunogenicity were assessed by the seroconversion rate of anti HPV6/11/16/18/33/45/52/58 neutralizing antibodies after day 31 post last dose, among the subjects who were aged 9-45 and seronegative before vaccination
Number of subjects receiving the 3-doses scheduled vaccination with antibody responses as assessed by IgG antibody GMT and seroconversion rate | day 31 post last dose
  Immunogenicity were assessed by the seroconversion rate and GMT of anti HPV6/11/16/18/33/45/52/58 IgG antibodies after day 31 post last dose, among the subjects who were aged 9-45 and seronegative before vaccination
The immunogenicity of subjects receiving 3 doses of vaccination was assessed by IgG antibodies and neutralizing antibodies | day 31 post last dose
  Immunogenicity were assessed by the seroconversion rate and GMT (4-fold increase rate) of anti HPV6/11/16/18/33/45/52/58 IgG and neutralizing antibodies after day 31 post last dose, among the subjects who were aged 9-45 and seropositive before vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Ting Huang, Study Director — Sichuan Provincial Center for Disease Control and Prevention
Locations (1):
- Center for Disease Control and Prevention, Mianzhu, Sichuan, China